CLINICAL TRIAL: NCT06911541
Title: Clinical Validation of a Novel, Accelerometer Based, Continuous Respiratory Rate Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eupnea AS (Industry)
Collaborators: Haraldsplass Deaconess Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Eupnea-2025-01
Record Dates: First submitted 2025-02-13; First posted 2025-04-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Rate Accuracy Test; Capnography; Wireless Vital Signs Monitoring System; Respiratory Rate
Keywords: Respiratory rate; wireless monitoring; accelerometer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult hospitalized patients (Experimental): Patients are being monitored for one hour with a wireless, accelerometer based respiratory rate sensor and a capnograph.
  Interventions: Device: Wireless respiratory rate monitor

INTERVENTIONS:
Device: Wireless respiratory rate monitor — This sensor is being fasten on the chest of the patients and measures respiratory rate with the help of an accelerometer. Data is being sent wireless to a backend monitor.

SUMMARY:
Comparing a wireless accelerometer-based sensor that continuously measure breathing rate with the gold standard capnography. The aim is to evaluate if both methods are equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Hospital
* Expected to remain undisturbed for at least one hour

Exclusion Criteria:

* Not able to give informed consent
* Use of high flow oxygen therapy
* Skin disease preventing proper attachment of the sensor
* Implanted electronic medical device.
* Known infection or colonisation with microbes necessitating protective measures above routine care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Validation of correctness of the sensor | one hour
  The respiratory rate measured by the sensor is being compared to the respiratory rate by capnography. A discrepancy of +- 3 breaths/min is within the acceptable range.

CONTACTS AND LOCATIONS:
Locations (1):
- Haraldsplass Deaconess Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Steihaug OM, Sjoset TE, Stordal AS, Sleire AD, Odegaard-Olsen O, Tunset A, Jammer I. Clinical validation of a novel accelerometer-based respiratory rate monitor. J Clin Monit Comput. 2026 Feb 7. doi: 10.1007/s10877-026-01419-x. Online ahead of print. PMID 41649789